CLINICAL TRIAL: NCT05558852
Title: Laparoscopic Central and Anterior Compartment Prolapse Surgery: A Meshless Sacrocolpopexy Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Resul Karakuş, Principle Investigator, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 84/2022
Record Dates: First submitted 2022-09-25; First posted 2022-09-28 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Prolapse Uterovaginal; Prolapse Bladder; Laparoscopy
Keywords: Laparoscopy; Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: Anticipated 25 patients will be evaluated and operated with meshless method.
Masking Description: Only one attending surgeon will operate the all participants. The patients will be evaluated pre-operatively by the surgeon and postoperatively 6th months by a different physician ( who is practicing as a gynecologist in the same hospital).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meshless Approach (Experimental): Laparoscopic Sacrocolpopexy in central or anterior compartment prolapse.
  Interventions: Procedure: Laparoscopic Meshless Sacrocolpopexy Technique

INTERVENTIONS:
Procedure: Laparoscopic Meshless Sacrocolpopexy Technique — Meshless sacrocolpopexy: laparoscopic approach to central and anterior compartment prolapse

SUMMARY:
Mesh is widely applied in the abdominal approach to pelvic organ prolapse surgery, and sacrocolpopexy-sacrohysteropexy is the gold standard application, particularly for central compartment abnormalities. There are numerous disadvantages associated with the use of mesh. In some studies, the rate of mesh complications (such as mesh erosion, contraction, response, and pain) can reach 20%. This surgical approach aims to provide laparoscopic repair of pelvic organ prolapse without the use of mesh, hence avoiding the difficulties associated with mesh.

DETAILED DESCRIPTION:
Patients who present to the Zeynep Kamil Education and Research Hospital Gynecology and Obstetrics Clinic between July 2022 and April 2023 with the complaint of prolapse and have uterine or vaginal cuff prolapse due to a central defect or cystocele due to an anterior compartment defect and are indicated for surgery will be included in the study.The surgeries will be performed laparoscopically after obtaining their written consent.

The Technique;

1. The anterior promontory and the presacral area are dissected to expose the anterior longitudinal ligament.
2. Dissection from this region, extension of the right sacrouter ligament from the lateral to the vaginal cuff or retrocervical region as well as visualization of the right ureter, isolation of the right sacrouterine ligament.
3. Dissection of the vesicovaginal space by cutting the vesicouterine peritoneum and eradication of the bladder. Lower limit of anterior compartment dissection; Exposing the puboservicovaginal fascia sufficiently to repair the anterior defect and exposing the defect.
4. Dissection of the Yabuki space to control the entrance of the ureters into the bladder during anterior compartment dissection.
5. Performing a hysterectomy and suturing the vaginal cup if additional gynecological indications are present. (in women with a uterus).
6. Repairing the defective pubocervico-vaginal fascia using 2.0 prolene for an anterior compartment defect and suturing this fascia to the cervical ring or sacrouterine ligaments in the vaginal cuff using 2.0 prolene.
7. Attaining the sacral promontory with two strong sutures starting from the vaginal cuff or cervix using 1.0 prolene and continuous circular sutures along the right sacrouterine ligament while using the same suture.
8. After passing 1 strong suture through the anterior longitudinal ligament, the same suture will be continued along the right sacrouterine ligament in a continuous and circular manner.
9. Knotting where the suture begins to create sufficient tension (maintaining the vaginal cuff level at -2) (The sacrocolpopexy technique: transforming the sacrouterine ligament into a rope with an insoluble suture material).
10. Finally, providing peritonization with 2.0 vicryl and, if indicated, culdoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Female patients older than 30 years and younger than 80 years old
* Patients who provided written consent for this surgical procedure

Exclusion Criteria:

* Patients who cannot obtain anesthesia approval for laparoscopic surgery
* Patients with asymptomatic pelvic organ prolapse
* Patients with active pelvic inflammatory disease
* Patients who have a confirmed or suspected pregnancy or malignancy
* Patients who have an unexplored abnormal cervical-uterine cytology

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients in between 30 to 80 years old with a symptomatic vaginal cuff/uterine prolapse and/or cyctocele
Enrollment: 25 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
Visual analog Scale | 6 months after the operation
  Pain Scale of 0 to 10, aiming that the operation itself leaves no pain.
POP-Q classification | 6 months after the operation
  examination of pelvis organs, aiming that the vaginal cuff stays at -2 level and no recur.
PQOL | 6 months after the operation
  Aiming to see the increased quality of life by the questionnaire which is given preoperatively and postoperative 6th month.
FSFI | 6 months after the operation
  Aiming to see the increased quality of sexual life by the questionnaire which is given preoperatively and postoperative 6th month.
Urinary Incontinance | 6 months after the operation
  Questioning and examining patient after surgery related to urinary incontinancy complaint, and evaluating the incontinancy state with questionnaires of Incontinence Impact Questionnaire (IIQ-7) and Urinary Distress Inventory (UDI-6)

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil Maternity and Childrens Training and Research Hospital, Istanbul, Turkey (Türkiye)